CLINICAL TRIAL: NCT04004884
Title: Liver Safety Assessment During Ulipristal Acetate Treatment for Uterine Fibroids
Brief Title: Liver Safety Assessment During Ulipristal Acetate Treatment for Uterine Fibroids (LISA)
Acronym: LISA
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ULI-2019-05
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2019-07

CONDITIONS: Leiomyoma, Uterine; Liver Injury; Treatment Side Effects
Keywords: Ulipristal Acetate; Selective Progesterone Receptor Modulators; Leiomyoma; Liver injury
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UPA Treatment: Women who had completed a full 12-week treatment course of Ulipristal Acetate for symptomatic uterine fibroids since September 2018
  Interventions: Drug: Ulipristal Acetate

INTERVENTIONS:
Drug: Ulipristal Acetate — Assess the variations of liver blood test parameters during UPA treatment for symptomatic uterine fibroids
  Other Names: Esmya

SUMMARY:
Uterine fibroids are are the most common gynecological tumor. Among the pharmacological treatment options, ulipristal acetate (UPA) has proven to be effective in control of bleeding and reduction of size of fibroids.

Due to the appearance of some cases of subacute severe hepatic insufficiency in patients undergoing UPA treatment and the possible idiosyncratic effect of the drug, the European Medicine Agency (EMA) recommended performing liver function tests before, during and after each UPA treatment course as a minimization risk strategy to prevent drug induced liver injury (DILI).

The aim of the present study is to evaluate whether changes in transaminase levels or other DILI markers occur in patients receiving UPA in our center.

DETAILED DESCRIPTION:
INTRODUCTION Fibroids are benign monoclonal tumors originated from genetically predisposed uterine smooth muscular cells in a proper hormonal environment. Fibroid growth is dependent on the ovarian steroids estrogen and progesterone. In vivo models have shown that progesterone and the presence of its receptor are the main key points for fibroid growth, being PR stimulation the primary action of estrogens.

Multiple treatment options are currently available, including surgery (hysterectomy or myomectomy), uterine artery embolization, cryomyolysis, radiofrequency myolysis, high-intensity focused ultrasound, and pharmacological treatment. Proper counseling about all therapeutic approaches should be discussed with the patient, explaining pros and cons of every treatment and taking into consideration several clinical factors such as number, location and fibroid size, age and desire for future pregnancies. Final decision of the best treatment should be taken according to the patient's desire.

Uterine fibroids still represent the most frequent indication for hysterectomy, which associates a low but significant risk of vascular, intestinal and urinary complications. Non-surgical treatments represent a good option for those young patients in order to avoid surgical scars on uterine surface and the risk of hysterectomy. Due to the Es and Prog dependent status, fibroid-related symptoms often cease once menopause status is achieved, so selected perimenopausal patients could also benefit from those therapies and avoid a surgery.

Among the pharmacological treatment options, gonadotropin-releasing hormone agonists (GnRHa) are effective in reducing bleeding and uterine volume, but with considerable side-effects due to the estrogen-suppression status. Ulipristal acetate (UPA) have been shown to be effective in bleeding control, induction of amenorrhea and fibroid reduction when compared to GnRHa, with fewer side effects as it maintains estradiol at mid-follicular phase levels. Pre-surgical UPA treatment allows recovery of Hb levels and reduction in fibroid size, allowing better minimally invasive surgery procedures. On selected patients, long-term intermittent treatment with UPA offers an alternative to surgery allowing patients to reach menopause status without surgery.

In February 2018, the European Medicines Agency (EMA) announced temporary restrictive measures to UPA treatment as 8 cases of severe liver injury were potentially linked to UPA administration. After the Pharmacovigilance Risk Assessment Committee (PRAC) evaluation concluded, the association between UPA and drug induced liver injury (DILI) was neither confirmed nor excluded. As a conclusion, the EMA stated that the benefits of UPA for the treatment of symptomatic uterine fibroids clearly outweigh the risks, but risk-minimization measures were needed in order to avoid the rare but serious possible liver injury.

In this work, the investigators evaluated evaluate whether changes in transaminase levels or other DILI markers occur in patients receiving UPA in the study center.

MATERIAL AND METHODS Retrospective observational study to assess the variations of liver blood test parameters during UPA treatment for symptomatic uterine fibroids. The study is approved by the ethics committee of the study site and will be conducted in accordance with the principles of the International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines Investigators will include all women who had completed a full 12-week treatment course of UPA for symptomatic uterine fibroids since September 2018. All patients will provide written informed consent. As stated by EMA recommendations, all patients will perform a blood test including liver parameters (AST, ALT, AF, GGT, bilirubin) before initiating the treatment, monthly during the 12-week treatment course, and an additional test 2-4 weeks after ending treatment. All data will be collected in an anonymized database with restricted access to investigators

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Symptomatic uterine fibroids
* Being prescribed UPA as a treatment for symptomatic uterine fibroids according to regular practice.

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Previous or active hepatic disease
* Transaminase (AST,ALT) blood levels higher than 3 times the upper normal limit.
* Bilirubin blood levels higher than 3 times the upper normal limit.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women who had completed a full 12-week treatment course of UPA for symptomatic uterine fibroids since September 2018.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Transaminase levels | 12 weeks
  Variations on AST or ALT blood levels during UPA treatment course.

SECONDARY OUTCOMES:
Gamma Glutamyl Transferase (GGT) levels | 12 weeks
  Variations on GGT blood levels during UPA treatment course.
Bilirubin levels | 12 weeks
  Variations on bilirubin blood levels during UPA treatment course.
Alkaline phosphatase (AF) levels | 12 weeks
  Variations on AF blood levels during UPA treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Estadella, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided